CLINICAL TRIAL: NCT05597371
Title: An Analysis of Changes in the Use of Telecommunication Platform in National Taiwan University Hospital During the Time of Global COVID-19 Pandemic
Brief Title: An Analysis in the Use of Telecommunication Platform
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202107160RINC
Record Dates: First submitted 2022-10-20; First posted 2022-10-28 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: the Use of the Platform

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: the use of the platform — the use of the platform

SUMMARY:
The COVID-19 pandemic becomes a global challenge. Beneficial to being an island country and having appropriate policies, there were only few imported cases in Taiwan. However, many locally acquired cases came out in the mid of this May. The hospital policy about containing infection changed accordingly.

A real-time communication platform for the health care workers was designed and embedded in the hospital information system of the emergency department in 2018. The functions included sending messages to certain staff, pop-up reminders, and tracking messages. This study aims to evaluate the use of the communication platform during the COVID pandemic.

DETAILED DESCRIPTION:
The COVID-19 pandemic becomes a global challenge. Beneficial to being an island country and having appropriate policies, there were only few imported cases in Taiwan. However, many locally acquired cases came out in the mid of this May. The hospital policy about containing infection changed accordingly.

A real-time communication platform for the health care workers was designed and embedded in the hospital information system of the emergency department in 2018. The functions included sending messages to certain staff, pop-up reminders, and tracking messages. This study aims to evaluate the use of the communication platform during the COVID pandemic.

ELIGIBILITY:
Inclusion Criteria:

healthcare workers with using the communication platform.

Exclusion Criteria:

healthcare workers without using the communication platform.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: ED visits of the emergency department of the National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 1000000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
the number of the use of the communication platform during the COVID pandemic | from 2018 to 2022
  the number of the use was divided by the visits

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ching Lien, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Department of Emergency Medicine, National Taiwan University Hospital, Taipei, Taiwan